CLINICAL TRIAL: NCT01679457
Title: Assessing Models of Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Utah State University (Other)
Responsible Party: Principal Investigator, Nate Gruner, Staff Behavior Therapist, Mclean Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-P-001010/1; McLean
Record Dates: First submitted 2012-08-22; First posted 2012-09-06 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Obsessive-compulsive Disorders and Symptoms
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT-Focused ERP (Experimental): One Session.
  Interventions: Behavioral: TAU-ERP
- TAU-ERP (Active Comparator): One Session.
  Interventions: Behavioral: ACT-Focused ERP

INTERVENTIONS:
Behavioral: ACT-Focused ERP
  Arms: TAU-ERP
Behavioral: TAU-ERP
  Arms: ACT-Focused ERP

SUMMARY:
The objective of this study is to learn how to improve treatment for clients who are working hard in treatment at the McLean Hospital Obsessive Compulsive Disorder Institute (OCDI), but who are not making the progress that would typically be expected. Therefore, the investigators will be comparing the performance of such clients in a treatment as usual (TAU)-Exposure and Response Prevention (ERP) session with their performance in an Acceptance and Commitment Therapy (ACT)-focused ERP session that follows an ACT booster session. The investigators hypothesize that clients will perform significantly better in the ACT-focused ERP session than they will in the TAU-ERP session. More specifically, the investigators hypothesize that clients and an independent rater will report that in the ACT-focused ERP session, clients performed significantly fewer rituals and/or avoidance behaviors, experienced comparable levels of distress, exerted significantly more effort, had significantly less difficulty getting started with the ERP, were significantly less influenced by their uncomfortable thoughts/feelings, were significantly more willing to experience discomfort, were significantly more focused on working towards what is important to the client. The investigators also hypothesize that an independent rater will rate clients as significantly more compliant with the ACT-focused ERP session than with the TAU-ERP session. The investigators also hypothesize that clients will rate the ACT-focused ERP session as significantly more preferable and acceptable than the TAU-ERP session, and that they will report being significantly more willing to do the ACT-focused ERP session again.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults at least 18 years of age currently enrolled in the residential or day treatment program at the OCDI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Client Post-ERP Session Questions (Day 1). | Client Post-ERP Session Questions (Day 1) will be administered immediately after the "Day 1" TAU-ERP session.
Client Post-ERP Session Questions (Day 2). | Client Post-ERP Session Questions (Day 2) will be administered immediately after the "Day 2" ACT-focused ERP session.

CONTACTS AND LOCATIONS:
Overall Officials: Nate G Gruner, LICSW, Principal Investigator — Mclean Hospital
Locations (1):
- Obsessive Compulsive Disorder Institute at McLean Hospital, Belmont, Massachusetts, United States